CLINICAL TRIAL: NCT00142688
Title: Examining Psychosocial Mediators of Exercise Behavior
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 253; R01HL072947 (NIH); A04-102 (Other: HealthPartners Institute)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases | interventions — Exercise; Health

ARMS (2):
- 1 (Experimental): Tailored print-based intervention in which participants complete questionnaires and receive tailored feedback based on responses to the questionnaires. The intervention is delivered monthly during the first month, bi-monthly during months 2 and 3, and monthly during months 4-6. The intervention is completed through the mail.
  Interventions: Behavioral: Physical activity
- 2 (Active Comparator): Participants receive wellness materials delivered through the mail on the same schedule as the experimental condition. Physical activity materials are given to this group upon completion of the study.
  Interventions: Behavioral: Wellness

INTERVENTIONS:
Behavioral: Physical activity — Tailored print-based intervention in which participants complete questionnaires and receive tailored feedback based on responses to the questionnaires. The intervention is delivered monthly during the first month, bi-monthly during months 2 and 3, and monthly during months 4-6. The intervention is completed through the mail.
  Arms: 1
Behavioral: Wellness — Participants receive wellness materials delivered through the mail on the same schedule as the experimental condition. Physical activity materials are given to this group upon completion of the study.
  Arms: 2

SUMMARY:
The purpose of this study is to examine psychosocial mediators of exercise behavior.

DETAILED DESCRIPTION:
BACKGROUND:

Physical inactivity is related to many health problems, including increased risk of cardiovascular disease, hypertension, and cancer. Despite the health consequences of a sedentary lifestyle, only 25 percent of Americans meet the recommended levels of physical activity. Researchers postulate that theory-based interventions effectively influence physical activity behavior by changing theoretical constructs believed to be important for behavior change (i.e., potential mediators), such as self-efficacy (i.e., confidence in one's ability to be physically active). Unfortunately, previous studies have generally failed to adequately test the mediating effect of theoretical constructs using appropriate statistical mediator analyses as recommended by leading behavioral scientists and statisticians.

DESIGN NARRATIVE:

The study will examine the mediating effect of theoretical constructs based on the Transtheoretical Model (TTM) and Social Cognitive Theory (SCT). The study will address the methodological, measurement, and statistical limitations of previous studies. The investigators will randomly assign 420 healthy sedentary individuals to either a theory-based physical activity intervention or a contact control group. Physical activity behavior and the potential mediators will be assessed monthly over 12 months. They hypothesize that constructs based on the TTM and SCT (i.e., behavioral processes, cognitive processes, self-efficacy, and decisional balance) will mediate the relationship between group assignment (intervention vs. contact control) and physical activity behavior, such that the effect of the intervention on physical activity behavior relative to the contact control group will be attenuated when controlling for the mediators. They will also examine the importance of particular mediators for different population groups (e.g., age, gender), which will help to create more effective interventions for these groups. Finally, they will conduct a cost analysis to not only inform policy makers of the cost of delivering the intervention within our study but also to estimate the cost of delivering each component of the intervention (i.e., mediator). The analysis will estimate the cost of future refined interventions that incorporate those active components that affect the mediators and physical activity in this study. In summary, the study will identify which mediators (i.e., theoretical constructs) are most effective for increasing physical activity, which will have an important public health impact given that this will likely lead to more efficacious and less costly interventions.

ELIGIBILITY:
Inclusion Criteria:

* In good health
* Living a sedentary lifestyle

Max Age: 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2004-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Physical activity | Measured at baseline, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Lewis, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Lewis BA, Williams DM, Martinson BC, Dunsiger S, Marcus BH. Healthy for life: a randomized trial examining physical activity outcomes and psychosocial mediators. Ann Behav Med. 2013 Apr;45(2):203-12. doi: 10.1007/s12160-012-9439-5. PMID 23229158
- [Derived] Lewis BA, Williams DM, Frayeh A, Marcus BH. Self-efficacy versus perceived enjoyment as predictors of physical activity behaviour. Psychol Health. 2016;31(4):456-69. doi: 10.1080/08870446.2015.1111372. Epub 2015 Nov 18. PMID 26541890